CLINICAL TRIAL: NCT01468298
Title: Comparing the Global Posture Reeducation With Isostretching in Chronic Low Back Pain Patients
Brief Title: Global Posture Reeducation (GPR) Compared To Isostretching in Chronic Low Back Pain Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Universitario de Maringa (Other)
Responsible Party: Principal Investigator, Ligia Maria Facci, Principal Investigator, Clinical Professor, Centro Universitario de Maringa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 249/2010
Record Dates: First submitted 2011-10-25; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-10

CONDITIONS: Low Back Pain
Keywords: back pain; physical therapy; spine; rehabilitation; exercise
MeSH Terms: conditions — Low Back Pain; Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isostretching (Active Comparator)
  Interventions: Other: Isostretching
- Global Posture Reeducation (Active Comparator)
  Interventions: Other: Global Posture Reeducation

INTERVENTIONS:
Other: Isostretching — All of patients were accompanied by an individual treatment program composed by 12 sessions of 45 minutes, twice a week. The Isostretching method includes therapeutic different postures, lying, sitting or standing, and the positions were selected according to the postural changes of each patient, identified in the assessment. The Isostretching protocol involves nine positions held for a period of nine breaths, and every three cycles, the patient should rest for a period. The physical therapist used verbal commands to emphasize pursed lip breathing, self growth, curvatures correction and isometric of abdominal, paravertebral, quadriceps and gluteal muscles with the aim of optimizing the stretching and discouraging compensatory movements.
  Other Names: postural reeducation
  Arms: Isostretching
Other: Global Posture Reeducation — All patients were accompanied by an individual treatment program composed by 12 sessions of 45 minutes, twice a week, involving a series of active gentle movements and postures aimed at realigning joints, stretching shortened muscles and enhancing the contraction of antagonist muscles, thus avoiding postural asymmetry. The positions were selected according to the postural changes of each patient, identified in the assessment and these therapeutic postures imply an active involvement of the patient. The protocol includes three therapeutic postures, lying, sitting or standing, to be held for 15 minutes each. The physical therapist used verbal commands and manual contact to maintain the alignment and make the necessary postural corrections, with the aim of discouraging compensatory movements.
  Other Names: postural reeducation
  Arms: Global Posture Reeducation

SUMMARY:
The aim of this study was to investigate the changes in posture, flexibility, muscle strength, functional capacity, heart rate(HR), peripheral oxygen saturation, systolic blood pressure, diastolic blood pressure and intensity of pain in chronic low back pain underwent to Isostretching and GPR.

DETAILED DESCRIPTION:
It was selected 40 patients, from 40 to 59 years old, with chronic low back pain from CESUMAR Physiotherapy Clinic-Schoo. These were evaluated before and after treatment regarding posture by SAPO computer program; flexibility for lumbar Schober testing, sit and reach; muscle strength by dynamometry for trunk extensors and the maximum repetition test in a minute to abdominal and trunk extensors; functional capacity by Rolland-Morris Questionnaire; pain by visual analog scale; heart rate(HR) by polar frequencymetric; peripheral oxygen saturation by Finger Pulse Oximeter; and systolic and diastolic blood pressure with a Sphygmomanometer. The sample was divided in two groups (1-GPR with 11 patients, 2-Isostretching with 10 patients). All patients were accompanied by an individual treatment program composed by 12 sessions of 45 minutes, twice a week. It was considered statistically significant p values <0.05 obtained from the Student's t test.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-specific LBP in its chronic phase (pain lasting more than 12 weeks), from 40 to 60 years old.

Exclusion Criteria:

* scheduling conflicts
* lack of transportation
* disease that compromises their health during the treatment
* uncontrolled hypertension
* fibromyalgia
* history of spinal surgery in the last six months
* patients with neurological diseases
* individuals who demonstrate inability to understand or physical restraint for the exercises.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
functional capacity | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  Low back patients functional capacity were evaluated before and after 10 sesssions treatment regarding by Rolland-Morris Questionnaire.

SECONDARY OUTCOMES:
Posture | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  Posture were evaluated before and after 10 sessions treatment regarding posture by computer SAPO (Softwere Avaluation Posture Online) program.
flexibility | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  These were evaluated before and after 10 sessions treatment regarding posture, flexibility for lumbar Schober testing and sit and reach.
muscle strength | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  These were evaluated before and after 10 sessions treatment regarding muscle strength by dynamometry for trunk extensors and the maximum repetition test in a minute to abdominal and trunk extensors.
heart rate(HR) | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  It was measured heart rate (HR)by polar frequencymetric at start and for every 15 minutes in 10 sessions therapy.
peripheral oxygen saturation | Before and after 10 sessions and for every 15 minutes in therapyPatients will be followed for the duration of 10 sessions, an expected average of 5 weeks..
  It was measured peripheral oxygen saturation (SpO2) by Finger Pulse Oximeter at start and for every 15 minutes in therapy.
systolic blood pressure | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks..
  It was measured systolic blood pressure (SBP) with a Sphygmomanometer at start and for every 15 minutes in 10 sessions therapy. Blood pressure measurement was obtained by arterial occlusion by inflation of the cuff, correlating to the auscultation of the heartbeat with the values recorded in the column of mercury. The sounds perceived during the blood pressure measurement procedure are called Korotkoff sounds, and classified into five phases, with phase 1 (first sound) corresponding to the value of systolic blood pressure (SBP).
diastolic blood pressure | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  It was measured diastolic blood pressure (DBP) with a Sphygmomanometer at start and for every 15 minutes in 10 sessions therapy.Blood Ppressure measurement was obtained by arterial occlusion by inflation of the cuff, correlating to the auscultation of the heartbeat with the values recorded in the column of mercury. The sounds perceived during the blood pressure measurement procedure are called Korotkoff sounds, and classified into five phases, with phase 5 (muffling or disappearance of sound) corresponding value of diastolic blood pressure (DBP).
Intensity of Pain | Patients will be followed for the duration of 10 sessions, an expected average of 5 weeks.
  The low back intensity of pain were evaluated before and after 10 sessions treatment regarding pain by visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ligia M Facci, doctor, Principal Investigator — Centro Universitario de Maringa
Locations (1):
- Centro Universitário de Maringá, Maringá, Paraná, Brazil